CLINICAL TRIAL: NCT06792851
Title: ECHO-012 Kosmos Bladder Clinical Validation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EchoNous Inc. (Industry)
Collaborators: Rainier Clinical Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ECHO-012
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Bladder Disease; Bladder Retention Volume; Bladder Dysfunction; Bladder Function
MeSH Terms: conditions — Urinary Bladder Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Bladder Volume Measurement (Experimental): Pre- and post-void bladder volume assessment using Kosmos device by both nurse and sonographer and void volume measurement.
  Interventions: Device: Kosmos Bladder Volume Algorithm

INTERVENTIONS:
Device: Kosmos Bladder Volume Algorithm — Participants underwent Kosmos bladder volume assessment by both a nurse and an abdominal sonographer pre-void. Participants voided and measured void volume. Participants underwent Kosmos bladder volume assessment by both a nurse and an abdominal sonographer post-void. Kosmos calculated volume measurements were compared to volume measurements calculated using calipers placed by sonographers by hand.

SUMMARY:
The goal of this clinical trial is to compare the Kosmos Automatic Bladder Volume to the manual annotated bladder volume in participants across gender (male and female), age (children ages 7-17 and adults 18-89), and BMI strata (low to normal and high BMI). The hypothesis it aims to evaluate is: The Pearson correlation coefficient between Kosmos estimated bladder volume and manually annotated bladder volume will yield more than 0.90.

Participants will:

* Have their full bladders scanned and bladder volume calculated using the Kosmos Ultrasound Diagnositic System by both a nurse and sonographer.
* Participants will void and measure their urine volume.
* Participants empty bladders will be scanned and bladder volume calculated using the Kosmos Ultrasound Diagnositic System again by both a nurse and sonographer.
* Three sonographers will manually annotate the pre- and post-void exam images for each patient to calculate the manually annotated bladder volume.

ELIGIBILITY:
Inclusion Criteria:

* Read and sign an English consent form, or assent form, in the case of a minor child
* Read and complete an English demographic and general health survey, or have an LAR complete it for them in the case of a minor child
* Give consent for participation, or assent in the case of a minor child
* Able and willing to comply with study requirements
* Follow fluid consumption requirements prior to the study visit
* Those aged 7 years through 89 years, healthy as well as individuals with pelvic region abnormalities (if applicable), including but not limited to:

  i) Bladder cancer ii) Thickened bladder wall iii) Bladder stones iv) Current bladder or urinary tract infection

Exclusion Criteria:

* Adults over 89 years old
* Children under the age of 7
* Persons who are pregnant
* Persons who report an empty bladder upon arrival at their scheduled study visit
* Children in foster care, as a foster parent may not legally consent for a foster child
* Those who cannot or refuse to sign their consent or assent (including those with an LAR willing to provide consent)
* Those who cannot provide informed consent or whose LAR cannot provide consent
* Those who cannot speak or read English
* Participants from ECHO-010 Bladder AI Training and Validation Data Collection Study

Ages: 7 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Manual Bladder Volume vs. Kosmos Automated Bladder Volume | Post data acquisition (one month)
  Kosmos Automated Bladder Volume and exam images will be captured using the Kosmos Ultrasound Diagnostic System by a nurse and a sonographer for each participant with both a full and empty bladder. Three independent sonographers will manually measure exam images for bladder length (L), width (W), and height (H). Volume will be calculated using: Bladder Volume = k×L×D×W where k is the correction coefficient. These results from the three sonographers will be averaged. The Pearson correlation coefficient between the average manual bladder volume and the Kosmos calculated pre-void volume will be calculated using the following equation: r=[∑(x-xbar)(y-ybar)]/[∑(x-xbar)^2 ∑(y-ybar)^2] Where x is the manual bladder volume, y is the Kosmos bladder volume, xbar is the mean of the manual bladder volume, and ybar is the mean of the Kosmos bladder volume. A successful outcome would be a correlation coefficient (r) of >0.90 on bladder exams acquired by both nurses and sonographers.

CONTACTS AND LOCATIONS:
Overall Officials: Sheryl Marks, M.D., Principal Investigator — Rainier Clinical Research Center
Locations (1):
- Rainier Clinical Research Center, Renton, Washington, United States